CLINICAL TRIAL: NCT03962140
Title: Computed Tomography Assessment of Body Fat Distribution in Endometrial Cancer Patients
Brief Title: CT Assessment of BMI in Endometrial Cancer Patients
Status: Completed | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.RCHT.39
Record Dates: First submitted 2019-04-17; First posted 2019-05-23 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; CT-scan; Fat distribution; Obesity; Sarcopenia
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a retrospective study to investigate the association between body fat distribution and sarcopenia on CT-scan and oncological outcomes in endometrial cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of endometrial cancer
* Age: 18 years or older
* Abdominal CT-scan as part of pre-operative or post-operative staging work-up (<1 month after surgery)

Exclusion Criteria:

* Women with concurrent cancer
* Women with unknown body mass index

Ages: 18 Years to 99 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Endometrial cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The Investigation of Patients with High BMI and Survival Rates | 10 years
  To investigate the association between body fat distribution and sarcopenia on CT-scan and survival in endometrial cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom